CLINICAL TRIAL: NCT02317302
Title: FDG Tumor Heterogeneity During Chemoradiation as a Predictor of Response to Concurrent Radiation Therapy and Chemotherapy in Patients With Cervical Cancer
Brief Title: FDG Tumor Heterogeneity During Chemoradiation as a Predictor of Response in Patients With Cervical Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 201104322
Record Dates: First submitted 2014-12-10; First posted 2014-12-16 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Cervical Cancer; Uterine Cervical Cancer; Uterine Cervical Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- FDG-PET/CT or FDG-PET/MR (Experimental): * Standard of care FDG-PET/CT or FDG-PET/MR at baseline
  * FDG-PET/CT or FDG-PET/MR after the 2nd but before the 3rd brachytherapy treatment
  * Standard of care 3 month post treatment FDG-PET/CT or FDG-PET/MR
  * We will perform the research-related FDG-PET on the PET/MR rather than the PET/CT if the patient is safe to undergo MR and agrees to undergo MR.
  * The standard of care imaging may be performed on the PET/CT scanner or the PET/MR scanner.
  Interventions: Device: FDG-PET/MR; Device: FDG-PET/CT

INTERVENTIONS:
Device: FDG-PET/MR
  Other Names: PET/MR
Device: FDG-PET/CT
  Other Names: PET/CT

SUMMARY:
In this study, 50 evaluable patients will undergo one FDG-PET study during their chemoradiation, in addition to the standard of care pretreatment and 3-month post-treatment clinical FDG-PET/CT or FDG-PET/MR scans. From all FDG-PET studies, tumor volume, SUVmax, FDGhetero, and texture maps will be obtained. Evaluating the changes in tumor SUVmax and heterogeneity during treatment will aid in better understanding the role of these biological parameters in inadequate response to chemoradiation. Other researchers, using MRI imaging, have evaluated changes in the cervical tumor volume during treatment. The investigators expect there will be variation in how cervical tumors shrink and change during chemoradiation and therefore we are going to use multiple measures in addition to tumor volume to evaluate cervical tumor metabolic heterogeneity. Being able to predict at diagnosis the patients who are at higher risk for persistent disease following chemoradiation would allow for future studies where these high risk patients could be specifically targeted with more aggressive therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have biopsy-proven cervical cancer (FIGO stage-Ib2-IVb).
* Patient must be at least18 years of age.
* Patient must be planning to receive chemoradiation therapy with cisplatin.
* Patient must have non-pregnant status if a female of childbearing potential. Women who have had a tubal ligation at least 12 months prior to study entry or a hysterectomy will be considered NOT of childbearing potential. Postmenopausal women must have been amenorrheic for at least 12 consecutive months to be considered NOT of childbearing potential.
* Patient may have distant metastatic disease provided the estimated survival is at least 1 year.
* Patient's tumor(s) must be FDG avid on baseline standard of care FDG-PET/CT or PET/MR imaging that was performed at Barnes-Jewish Hospital Clinical PET Facility.
* Patient must be able and willing to give informed consent.
* If the patient will be scanned on the PET/MR for the mid-treatment scan, they must be determined to be safe for exposure to the magnetic field. This will be determined the day of imaging by the technologist with the use of a screening form. If a patient is not safe for the PET/MR scanner, their mid-treatment images will occur on the PET/CT scanner in the Center for Clinical Imaging Research.

Exclusion Criteria:

* Patient must have no other active cancer at the time of diagnosis of cervical cancer.
* Patient cannot have received treatment for any malignancy, with the exception of non-melanoma skin cancer, in the past 5 years.
* Patient must not be an uncontrolled diabetic with a glucose of ≥ 200mg/dl at the time of PET imaging.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-06-28 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
Change in FDG heterogeneity (Using texture analysis) | Up to 5 years
  Using texture analysis
Change in SUVmax (SUVmax - maximum standardized uptake value = is a marker of tumor glucose metabolism and reflects tumor aggressiveness) | Up to 5 years
  SUVmax - maximum standardized uptake value = is a marker of tumor glucose metabolism and reflects tumor aggressiveness.

SECONDARY OUTCOMES:
Response to therapy based on FDG heterogeneity | Up to 5 years
Response to therapy based on SUVmax | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Perry Grigsby, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu